CLINICAL TRIAL: NCT02235142
Title: Localised Cancer of Prostate and Androgen Deficiency.
Brief Title: Prostatic Cancer Versus Androgen Deficiency
Acronym: AndroCan
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hopital Foch (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2013/01; 2012-A01742-41 (Other: ANSM)
Record Dates: First submitted 2014-09-05; First posted 2014-09-09 (Estimated); Last update posted 2022-01-20 (Actual); Status verified 2022-01

CONDITIONS: Cancer of Prostate
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Blood Specimen Collection

ARMS (1):
- Localised prostat cancer and androgen deficiency (Experimental)
  Interventions: Other: Blood sample

INTERVENTIONS:
Other: Blood sample

SUMMARY:
Open study to make a comparison between hypogonadism and euogonadism patients regarding the severity of prostate cancer. The purpose of this study is to determine the importance of the relationship between the hormonal status and the type of the tumor at the time of surgical intervention as well as follow up of the patients.

ELIGIBILITY:
Inclusion Criteria:

* Male patients over than 18 years of age, with localized, stage I or II prostate cancer, not receiving local treatment (radiation, phototherapy, thermotherapy,…) or hormonal therapy, showing indication of radical prostatectomy.

Exclusion Criteria:

* Absence of radical prostatectomy indication
* Patient received local or hormonal therapy prior to surgery
* Patients already enrolled in other clinical study incompatible with the study
* Patients on a treatment which can affect hormonal level (Prednisone, Ketoconazole, Abiraterone, Finasteride, Dutasteride)

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1614 (Actual)
Dates: Start 2013-06-03 (Actual); Primary Completion 2016-06-27 (Actual); Study Completion 2021-12-22 (Actual)

PRIMARY OUTCOMES:
Testosteron Serum level | The day prior to surgery
Gleason score | 5 years

CONTACTS AND LOCATIONS:
Locations (8):
- France (6):
  - Clinique Saint Augustin, Bordeaux
  - Hôpitaux Civils de Colmar, Colmar
  - Hôpital Henri Mondor, Créteil
  - La Pitié-Salpêtrière (AP-HP), Paris
  - Institut Mutualiste Montsouris, Paris
  - Hôpital Foch, Suresnes, Île-de-France Region
- CHU Pointe à Pitre, Pointe-à-Pitre, Guadeloupe
- CHU Fort de France, Fort-de-France, Martinique

REFERENCES:
- [Derived] Pattou M, Neuzillet Y, Ghoneim T, Bosset PO, Vanalderverelt V, Bohin D, Lugagne PM, Soorojebally Y, Schneider M, Cathelineau X, Roupret M, Drouin SJ, Lebret T. Evaluating the Safety of Delaying Surgery Beyond 9 Months in Localized Prostate Cancer Patients: Results From a Prospective Study With Propensity Score Matching. Int J Urol. 2025 Sep;32(9):1243-1249. doi: 10.1111/iju.70142. Epub 2025 Jun 4. PMID 40462596
- [Derived] Neuzillet Y, Raynaud JP, Dreyfus JF, Radulescu C, Rouanne M, Schneider M, Krish S, Roupret M, Drouin SJ, Comperat E, Galiano M, Cathelineau X, Validire P, Molinie V, Fiet J, Giton F, Lebret T, Botto H. Aggressiveness of Localized Prostate Cancer: the Key Value of Testosterone Deficiency Evaluated by Both Total and Bioavailable Testosterone: AndroCan Study Results. Horm Cancer. 2019 Feb;10(1):36-44. doi: 10.1007/s12672-018-0351-8. Epub 2018 Oct 6. PMID 30293206